CLINICAL TRIAL: NCT04926597
Title: Effect of Continued Nutritional Support at Hospital Discharge on Mortality, Frailty, Functional Outcomes and Recovery Trial: The EFFORT II Project
Brief Title: Effect of Continued Nutritional Support at Hospital Discharge on Mortality, Frailty, Functional Outcomes and Recovery
Acronym: EFFORT II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipp Schuetz (Other)
Responsible Party: Sponsor-Investigator, Philipp Schuetz, Prof. Dr. med., Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-00278; ex20Schuetz
Record Dates: First submitted 2021-06-01; First posted 2021-06-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Malnutrition
Keywords: Nutritional Support; Oral Nutritional Supplements; Frailty; Mortality; Morbidity
MeSH Terms: conditions — Malnutrition; Frailty | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Pragmatic, single blinded, open label randomised-controlled trial
Who Masked: Outcomes Assessor
Masking Description: This trial is single blinded (regarding outcome assessment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: individualized nutritional support (Experimental): Intervention group patients will receive individualized nutritional support to reach energy and protein goals with the support of an experienced, unblinded dietician and with use of oral nutritional supplements (ONS) as needed
  Interventions: Dietary Supplement: nutritional supplement; Other: individualized nutritional guidelines
- Control group: general information on healthy food habits (Other): Control group patients will receive nutritional counselling (general information on healthy food habits) at discharge, but no nutritional support strategy will be used during follow-up
  Interventions: Other: general nutritional information

INTERVENTIONS:
Dietary Supplement: nutritional supplement — daily use of one or more specific oral nutritional supplement with high energy/protein content (i.e., Resource Ultra, Resource 2.0 (Fibre), Resource Ultra Fruit).
  Arms: Intervention group: individualized nutritional support
Other: individualized nutritional guidelines — nutritional plan supervised by an experienced study dietician based on the usual home nutrition with possibility to increase intake by adaptation to patient preferences, between meal snaking and food enrichment/fortification. Every 2-4 weeks phone call by unblinded study dietician to follow nutritional intervention.
  Arms: Intervention group: individualized nutritional support
Other: general nutritional information — general information about health food behavior upon hospital discharge
  Arms: Control group: general information on healthy food habits

SUMMARY:
This study is to compare the sustained post-discharge nutritional support to reach individual energy and protein goals to usual care home nutrition in medical patients at nutritional risk.

DETAILED DESCRIPTION:
Malnutrition is a strong and independent long-term risk factor for mortality, rehospitalisation and functional decline, particularly in the elderly, polymorbid medical patient population. The randomized-controlled Effect of early nutritional support on Frailty, Functional Outcomes and Recovery of malnourished medical inpatients Trial (EFFORT, Lancet 2019) included 2028 patients in eight Swiss hospitals and found that nutritional support during the inhospital stay reduces very efficiently the risk for complications and mortality with numbers needed to treat (NNT) of 23 and 37, respectively.

Yet, the nutritional intervention was not continued after hospital discharge of patients and long-term follow-up data of patients showed a lack of sustained effect of the initial nutritional support strategy. There is a current lack of trial data investigating whether long-term use of nutritional support has a sustained effect on clinical outcomes in this patient population. This study is to compare the continuous use of nutritional support with the use of approved oral nutritional supplements to reach protein and energy goals and to analyze whether medical patients at nutritional risk show a sustained benefit from long-term nutritional support after hospital discharge, and why and how nutritional support affects the course of disease from a mechanistic physio-pathological standpoint.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Adult (age ≥18 years), medical patients
* Nutritional risk screening using the Nutritional Risk Screening (NRS): total score ≥3 points consisting of ≥1 points for impairment of the nutritional status [weight loss >5% in 3 month or food intake of 50-75% in the last week before hospital admission] plus ≥1 for the severity of the disease (i.e., cancer, chronic kidney disease, chronic heart failure, COPD) and other chronic diseases according to the definition of the "National Center for Chronic Disease Prevention and Health Promotion": Chronic diseases are defined broadly as conditions that last 1 year or more and require ongoing medical attention or limit activities of daily living or both .

Exclusion Criteria:

* after surgery
* unable to ingest oral nutrition
* need for long-term nutrition,
* terminal condition
* acute pancreatitis or acute liver failure
* patients discharged to a nursing home
* patients unlikely to comply with nutritional support treatment (e.g., dementia)
* COVID-Hospitalisation requiring intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
time to death from any cause (i.e., all-cause mortality) | Enrollment to 3 years
  time to death from any cause (i.e., all-cause mortality)

SECONDARY OUTCOMES:
Time to non-elective hospital readmission after discharge from the index hospital stay | assessed from Day 0 (study enrolment), then every 6 month through phone calls up to end of trial (approx 3 years)]
  Time to non-elective hospital readmission after discharge from the index hospital stay
Time to the first major complication | assessed from Day 0 (study enrolment), then every 6 month through phone calls up to end of trial (approx 3 years)]
  time to the first major complication including death, bacterial infection with need for antibiotic treatment, major cardiovascular event (i.e., stroke, intracranial bleeding, cardiac arrest, myocardial infarction) or pulmonary embolism, acute renal failure, gastro-intestinal events (including hemorrhage, intestinal perforation, acute pancreatitis)
Changes in functional status measured by the Barthel's index | assessed from Day 0 (study enrolment), then every 6 month through phone calls up to end of trial (approx 3 years)]
  Changes in functional status measured by the Barthel's index (scores range from 0 to 100, with higher scores indicating better functional status)
Changes in quality of life measured with the European Quality of Life 5 Dimensions index (German Version, EQ-5D index) | assessed from Day 0 (study enrolment), then every 6 month through phone calls up to end of trial (approx 3 years)]
  Changes in quality of life measured with the European Quality of Life 5 Dimensions index (German Version, EQ-5D index values range from 0 to 1, with higher scores indicating better quality of life)
Changes in quality of life measured with the visual-analogue scale (EQ-5D VAS) | assessed from Day 0 (study enrolment), then every 6 month through phone calls up to end of trial (approx 3 years)]
  Changes in quality of life measured with the visual-analogue scale (EQ-5D VAS) (scores range from 0 to 100, with higher scores indicating better health status).

OTHER OUTCOMES:
Change in body weight | assessed from Day 0 (study enrolment), then at 3, 6 and 12 months by home visits
  Change in body weight
Change in calf circumference to assess muscle mass | assessed from Day 0 (study enrolment), then at 3, 6 and 12 months by home visits
  Change in calf circumference to assess muscle mass
Change in bioelectrical impedance analysis (BIA) to assess body composition | assessed from Day 0 (study enrolment), then at 3, 6 and 12 months by home visits
  Change in bioelectrical impedance analysis (BIA) to assess body composition
Change in hand grip by means of handgrip strength through dynamometry (North Coast Medical Exacta™ Hydraulic Hand Dynamometer) to assess muscle strength | assessed from Day 0 (study enrolment), then at 3, 6 and 12 months by home visits
  Change in hand grip by means of handgrip strength through dynamometry (North Coast Medical Exacta™ Hydraulic Hand Dynamometer) to assess muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Schuetz, Prof. Dr. med., Principal Investigator — Kantonsspital Aarau, University Department of Internal Medicine
Locations (18):
- Spain (6):
  - Hospital Universitari Vall Hebron de Barcelona, Barcelona
  - Hospital Universitario de Getafe, Getafe
  - Complejo AComplejo Asistencial Universitario de León, León
  - Hospital U. Gregorio Marañón de Madrid, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (12):
  - Spital Zofingen, Zofingen, Canton of Aargau
  - Spital Emmental Burgdorf, Burgdorf, Canton of Bern
  - Spital Thun, Thun, Canton of Bern
  - Spital Lachen, Lachen, Canton of Schwyz
  - Kantonsspital Münsterlingen, Münsterlingen, Thurgau
  - Kantonsspital Aarau, University Department of Internal Medicine, Aarau
  - Bern University Hospital, Department of General Internal Medicine, Bern
  - Kantonsspital Lucerne, Department of Internal Medicine, Lucerne
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Klinik Hirslanden Zürich, Zurich
  - Stadtspital Zürich, Zurich
  - Universitätsspital Zürich, Zurich